CLINICAL TRIAL: NCT03896737
Title: A Multicenter, Open Label, Randomized Phase II Study Comparing Daratumumab Combined With Bortezomib-Cyclophosphamide-dexamethasone (Dara-VCd) Versus the Association of Bortezomib-Thalidomide-dexamethasone (VTd) as Pre Transplant Induction and Post Transplant Consolidation, Both Followed by a Maintenance Phase With Ixazomib Alone or in Combination With Daratumumab, in Newly Diagnosed Multiple Myeloma (MM) Young Patients Eligible for Autologous Stem Cell Transplantation
Brief Title: Daratumumab-bortezomib-dexamethasone (Dara-VCd) vs Bortezomib-Thalidomide-Dexamethasone (VTd), Then Maintenance With Ixazomib (IXA) or IXA-Dara
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: EMN Trial Office S.r.l. Impresa Sociale (Other)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN18
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: diagnosis; elderly; autologous stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma; Disease | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Dara-VCD versus VTd
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dara-VCd (Experimental): treatment period includes administration of four 28-day cycles of induction with Dara- VCd; then patients will undergo transplant and finally they will receive two 28-day cycles of Dara-VCd consolidation treatment.
  The response will be assessed after each cycle. Patients in the first randomization will be stratified according to FISH (standard/missing vs high risk,defined as del17, t 4;14, t 14;16) and ISS (I vs II and III).
  TREATMENT SCHEMA - INDUCTION Daratumumab: 16 mg/Kg given by IV infusion on days 1, 8, 15, 22, on cycles 1-2 and on days 1, 15 on cycles 3-4.
  Bortezomib: 1.3 mg/m2 given SC injection on days 1, 8,15, 22; Cyclophosphamide: 300 mg/ m2 given orally or IV infusion on days 1, 8, 15, 22; Dexamethasone: 40 mg given orally or by IV infusion on days 1, 8, 15,22 Repeat for four 4-week induction cycles.
  Interventions: Drug: Daratumumab plus Velcade Cyclophosphamide Dexamethasone
- VTd (Active Comparator): treatment period includes administration of four 28-day cycles of induction with VTd; then patients will undergo transplant and finally they will receive two 28-day cycles of VTd consolidation treatment.
  TREATMENT SCHEMA INDUCTION
  ARM VTd:
  Bortezomib: 1.3 mg/m2 given by SC injection on days 1, 4, 8, 11 of 28-day cycle; Thalidomide: 100 mg given orally on days 1-28. Dexamethasone: 20 mg given orally or by IV injection on days 1, 2, 3, 4, 8, 9, 10 and 11 of every 28-day cycle.
  Repeat for four 4-week induction cycles.
  Interventions: Drug: Velcade Thalidomide Dexamethasone

INTERVENTIONS:
Drug: Daratumumab plus Velcade Cyclophosphamide Dexamethasone — To compare Dara-VCd versus VTd as pre transplant induction and post transplant consolidation, both followed by a maintenance phase with Ixazomib alone or in combination with Daratumumab, in newly diagnosed Multiple Myeloma (MM) young patients eligible for autologous stem cell transplantation.
  Arms: Dara-VCd
Drug: Velcade Thalidomide Dexamethasone — To compare Dara-VCd versus VTd as pre transplant induction and post transplant consolidation, both followed by a maintenance phase with Ixazomib alone or in combination with Daratumumab, in newly diagnosed Multiple Myeloma (MM) young patients eligible for autologous stem cell transplantation.
  Arms: VTd

SUMMARY:
This protocol is a phase II multicenter, randomized, open label study designed to assess the efficacy and safety of daratumumab combined with bortezomib, cyclophosphamide and dexamethasone (Dara-VCd) versus the association of bortezomib, thalidomide and dexamethasone (VTd) as pre transplant induction and post transplant consolidation, followed by maintenance with ixazomib alone or in combination with daratumumab, in newly diagnosed multiple myeloma (MM) patients eligible for autologous stem cell transplantation.

Patients enrolled in the Dara-VCd arm will receive: 4 cycles of daratumumab-bortezomib-cyclophosphamide-dexamethasone induction, followed by transplantation and 2 cycles of daratumumab-bortezomib-cyclophosphamide-dexamethasone consolidation. The choice of cyclophosphamide in combination with bortezomib and dexamethasone is suggested by the better safety profile of cyclophosphamide, in comparison with thalidomide and the efficacy of the alkylator agent, when combined with bortezomib.

Once-weekly bortezomib seems to be equally effective and better tolerated than the standard twice weekly schedule. The outcomes and response rate did not appear to be affected by the bortezomib dosing schedule.

Patients enrolled in the VTd arm will receive: 4 cycles of bortezomib-thalidomide-dexamethasone induction, followed by autologous transplantation and 2 cycles of bortezomib-thalidomide dexamethasone as consolidation. The VTd drug association is the current standard first line induction therapy for multiple myeloma patients who are eligible to stem cell transplantation.

At the end of consolidation phase patients with at least a partial response (≥ PR) will be rerandomized (assigned by chance) to one of 2 treatment groups to receive maintenance treatment with ixazomib alone or in combination with daratumumab. Patients will receive treatment until any sign of progression or intolerance, up to 24 months.

DETAILED DESCRIPTION:
INDUCTION AND CONSOLIDATION REGIMEN:

Arm Dara-VCd:

Daratumumab: 16 mg/Kg given by IV infusion on days 1, 8, 15, 22, on cycles 1-2 and on days 1, 15 on cycles 3-4.

Bortezomib: 1.3 mg/m2 given subcutaneous (SC) injection on days 1, 8,15, 22; Cyclophosphamide: 300 mg/ m2 given orally or by IV infusion on days 1, 8, 15, 22; Dexamethasone: 40 mg given orally or by IV infusion on days 1, 8, 15, 22 Repeat for four 4-week induction cycles. After induction all patients will be given Cyclophosphamide at the dose of 3 g/m2, followed by Granulocyte Colony-Stimulating Factor (G-CSF) for stem cell collection. Cyclophosphamide will start 4-6 weeks after start of the fourth cycle of therapy.

Stem cell collection will be performed as soon as CD34+ cells are present in peripheral blood, which is usually between 9-14 days after first day of Cyclophosphamide. Stem cells will be harvested at a minimum of 4 x 106 CD34+ cells/kg and cryopreserved. In case insufficient stem cells are collected the procedure may be repeated or alternatively bone marrow stem cell collection may be performed or Plerixafor may be used.

4-6 weeks after cyclophosphamide patients will be treated with High Dose Melphalan followed by autologous stem cell reinfusion according to the schedule below:

* Melphalan 200 mg/ m² day - 2 i.v. rapid infusion
* Stem cell infusion Minimum of 2 x 10^6CD34+cells/kg day 0 90-120 days after Melphalan administration consolidation treatment will be administered: Daratumumab: 16 mg/Kg given by IV infusion on days 1, 15; Bortezomib: 1.3 mg/m2 given by SC injection on days 1, 8, 15, 22; Cyclophosphamide: 300 mg/ m2 given orally or by IV infusion on days 1, 8, 15, 22; Dexamethasone: 40 mg given orally or by IV infusion on days 1, 8, 15, 22. Repeat for 2 4-week consolidation cycles.

Arm VTd:

Bortezomib: 1.3 mg/m2 given by SC injection on days 1, 4, 8, 11 of 28-day cycle; Thalidomide: 100 mg given orally on days 1-28. Dexamethasone: 20 mg given orally or by IV injection on days 1, 2, 3, 4, 8, 9, 10 and 11 of every 28-day cycle.

Repeat for 4 4-week induction cycles. After induction all patients will be given Cyclophosphamide at the dose of 3 g/m2, followed by G-CSF for stem cell collection. Cyclophosphamide will start 4-6 weeks after start of the fourth cycle of therapy.

Stem cell collection will be performed as soon as cluster of differentiation 34 (CD34)+ cells are present in peripheral blood, which is usually between 9-14 days after first day of Cyclophosphamide. Stem cells will be harvested at a minimum of 4 x 106 CD34+ cells/kg and cryopreserved. In case insufficient stem cells are collected the procedure may be repeated by using also Plerixafor or alternatively bone marrow stem cell collection may be performed.

4-6 weeks after cyclophosphamide patients will be treated with High Dose Melphalan followed by autologous stem cell reinfusion according to the schedule below:

* Melphalan 200 mg/ m² day -2 i.v. rapid infusion
* Stem cell infusion Minimum of 2 x 10^6CD34+cells/kg day 0 90-120 days after Melphalan administration consolidation treatment will be administered: Bortezomib: 1.3 mg/m2 given by SC injection on days 1, 4, 8, 11 of 28-day cycle; Thalidomide: 100 mg given orally on days 1-28; Dexamethasone: 20 mg given orally or by IV injection on days 1, 2, 3, 4, 8, 9, 10 and 11 of every 28-day cycle.

Repeat for 2 4-week consolidation cycles.

MAINTENANCE TREATMENT:

All patients in ≥ PR after consolidation will be randomized to receive:

Arm I Ixazomib 3 mg on days 1, 8, 15 of cycle 1-4, followed by ixazomib 4 mg on days 1, 8, 15 cycles from cycle 5*.

Repeat each cycle every 28 days. Patients will receive treatment until any sign of progression or intolerance, up to 24 months.

Arm II Ixazomib 3 mg on days 1, 8, 15 of cycle 1-4, followed by ixazomib 4 mg on days 1, 8, 15 cycles from cycle 5*.

Daratumumab 16 mg/kg on day 1. Repeat each cycle every 28 days. Patients will receive treatment until any sign of progression or intolerance, up to 24 months.

*The dose escalation is admitted only in case there have been no non-hematologic Adverse Events (AEs) ≥ Grade 2 related to study drug and no dose interruptions related to study drug toxicities.

Patients in the first randomization will be stratified according to fluorescent in situ hybridization (FISH) (standard/missing vs high risk, defined as del17, t 4;14, t 14;16) and International Staging System (ISS) (I vs II and III) Patients randomized to maintenance treatment will be stratified according to induction treatment and Minimal Residual Disease (MRD) status by nerve growth factor (NGF) (positive and not evaluable vs negative).

STATISTICAL DESIGN A total of 400 patients will be needed, in according to the study design, to provide a power of at least 85% to the statistical analysis with a two sided alpha error of 0.05 (see study protocol for details).

The statistical analysis will be performed in according to the intention to treat principle and will include summary of descriptive statistics (arithmetic mean and standard deviation, minimum and maximum, median with the interquartile range as appropriate) for continuous variables, absolute frequencies and percentages will be reported for qualitative variables. 95% Confidence intervals will be provided for variables subjected to statistical inference.

Proportions will be compared between treatment groups by use of the chi-square test or Fisher's exact test.

Kaplan-Meier method will be used for survival analyses to estimate and compare survival outcomes.

The log-rank test will be adopted to compare survival curves. Multivariable analysis, using semi parametric Cox proportional hazard regression model, will be performed to assess factors significantly affecting the progression free survival.

The safety analysis will include all patients randomized who will receive at least one dose of study treatment and the toxicity will be compared between treatment groups with chi-squared test.

All tests will be considered significant with p values less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age and ≤ 65 years.
* Patient eligible for autologous stem cell transplantation (ASCT).
* Left Ventricular Ejection Fraction (LVEF) ≥ 40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Multigated Acquisition Scan (MUGA) is acceptable if ECHO is not available.
* Newly diagnosed multiple myeloma patient.
* Patient has given voluntary written informed consent before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* Patient with documented multiple myeloma and measurable disease as defined by:
* Monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytoma
* Measurable disease as defined by at least one of the following:

  * serum M-protein level ≥1 g/dL or urine M-protein level ≥200 mg/24 hours; or
  * Light chain multiple myeloma: Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.
* Evidence of end organ damage/presence of biomarkers of malignancies, specifically:
* Hypercalcaemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11 mg/dL)
* Renal insufficiency: creatinine clearance (CLcr)<40 mL per minute (measured or estimated by validated equations) or serum creatinine >177 μmol/L (>2 mg/dL)
* Anaemia: haemoglobin value of >20 g/L below the lower limit of normal, or haemoglobin value <100 g/L
* Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT. If bone marrow has <10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement
* Any one or more of the following biomarkers of malignancy:
* Clonal bone marrow plasma cell percentage ≥ 60% (clonality should be established by showing κ/λ-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used)
* Involved:uninvolved serum free light chain ration ≥ 100 (values based on the serum Free light assay. The involved free light chain must be ≥100 mg/L)

  -> 1 focal lesion on MRI (magnetic resonance imaging) studies (each focal lesion must be 5 mm or more in size) Patient is, in the investigator(s) opinion willing and able to comply with the protocol requirements.
* Women of childbearing potential must commit to either abstain continuously from heterosexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [birth control pills, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin prior to dosing through 90 days after the last dose of study drug. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy.
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 90 days after the last dose of study drug.
* Patient with an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 or Karnofsky performance status ≥ 60%.
* Pretreatment clinical laboratory values within 30 days of enrolment:
* Platelet count ≥75 x 109/L;
* Absolute neutrophil count (ANC) ≥ 1 x 109/L (G-CSF use is permitted);
* Corrected serum calcium <14 mg/dL (<3.5 mmol/L);
* Aspartate transaminase (AST) ≤ 2.5 x the upper limit of normal (ULN);
* Alanine transaminase (ALT) ≤ 2.5 x the ULN;
* Total bilirubin ≤ 1.5 x the ULN;
* Calculated or measured creatinine clearance ≥ 30 mL/minute.
* Patient has a life-expectancy >3 months.

Exclusion Criteria:

* Patient with a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, smoldering MM or Plasma Cell Leukemia (PCL). Monoclonal gammopathy of undetermined significance is defined by presence of serum M-protein <3 g/dL, clonal bone marrow plasma cells <10%, and absence of end-organ damage or amyloidosis that can be attributed to the plasma cell proliferative disorder. Smoldering multiple myeloma is defined as serum monoclonal protein ≥ 30 g/L or urinary monoclonal protein ≥ 500 mg per 24 h and/or clonal bone marrow plasma cell 10-60% with absence of related organ or tissue impairment or end-organ damage or amyloidosis. Plasma cell leukemia is defined as presence of circulating plasmacells (PCs) >2×109/L in peripheral blood or a peripheral blood plasmacytosis >20%
* Patient with a diagnosis of Waldenström's disease, or other conditions in which immunoglobulin M (IgM) M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
* Patient has prior or current systemic therapy or SCT for multiple myeloma, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
* Patient has peripheral neuropathy of grade 2 or higher as defined by National Cancer Institute Common Toxicity Criteria (NCI CTC) 4.0.
* Patient is exhibiting clinical signs of meningeal involvement of multiple myeloma.
* Clinical active infectious hepatitis type A, B, C or HIV.
* Subject has known chronic obstructive pulmonary disease (COPD) (defined as a Forced Expiratory Volume In 1 second (FEV1) <60% of predicted normal), persistent asthma, or a history of asthma within the last 2 years. Subjects with known or suspected COPD or asthma must have a FEV1 test during screening.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations.
* Contraindication to any of the required concomitant drugs or supportive treatments.
* Pregnant or lactating females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 5 years
  PFS in part 1 and part 2 of the study will be measured from the date of first or second randomization to the date of first observation of disease progression or death to any cause as an event. Subjects who withdraw from the study will be considered censored at the time of the last complete disease assessment. Subjects who complete the study, have no progressed, and are still alive at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to followup prior to the end of the study have no progressed, and are still alive will also be censored at the time of last contact.
MRD negativity | 5 years
  MRD evaluation by clonotypic analysis of Immunoglobulin heavy chain (IgH) Variable-Diversity-Junctional (VDJ) gene rearrangement will be performed on bone marrow (BM) samples obtained by the end of induction and consolidation and thereafter every 6 mm after the first maintenance treatment dose. The Clonal Sequencing (ClonoSEQTM) assay (Adaptive Biotechnologies, Seattle) will be used at sensitivity thresholds of 10-3 (1 cancer cell per 1,000 nucleated cells), 10-4 and >/= 10-5. The rate of MRD negativity in each of the treatment arms of study protocol is determined as the proportion of patients with MRD negativity (>/=10-5 sensitivity level) at any established treatment point. Patients who withdraw from the study or are lost to Follow-up (FU) will be considered censored a t the time of the last MRD assessment. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 5 years
  ORR will include at least PR using the International Response Criteria reported by Durie et al. (Appendix V) Categories of response will include stringent Complete Response (sCR), CR, Very Good Partial Response (VGPR), PR, Stable Disease (SD) and PD. If, during the course of the study, other relevant categories are identified in the literature, then these categories may be added. Responders are defined as subjects with at least a PR.
Progression free survival 2 (PFS2) | 5 years
  PFS2 will be measured from the date of first randomization to the date of observation of second disease progression (i.e. progression after the second line of therapy) or death to any cause as an event. In case of date of second progression is not available, date of start of third line treatment can be used. Subjects who withdraw from the study will be considered at the time of the last complete disease assessment. Subjects who complete the study, have no progressed, and are still alive at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to follow-up prior to the end of the study have no progressed, and are still alive will also be censored at the time of last contact
Duration of response (DoR) | 5 years
  Time between first documentation of response and PD. Responders without disease progression will be censored either at the time of lost to follow-up, at the time of death due to other cause than PD, or at the end of the study.
Overall survival (OS): | 5 years
  OS is defined as the time between the date of first randomization and death. Subject who die, regardless the cause of death, will be uncensored as an event. Alive subjects who withdraw consent for study will be censored at the time of withdrawal. Subjects who complete the study and are still alive at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to follow-up prior to the end of the study will also be censored at the time of last contact.
Time to the next anti-myeloma therapy (TNT) | 5 years
  TNT will be measured from the date of first randomization to the date of next anti-myeloma therapy. Death due to disease progression before starting therapy or death of any causes, will be considered an event. Subjects who withdraw from the study will be considered censored at the time of the last complete disease assessment. Subject who complete the study, have no progressed, and are still alive at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to follow-up prior to the end of the study will also be censored at the time of last contact.
MRD by NGF and Positron Emission Tomography (PET)/CT | 5 years
  Immunophenotypic CR is defined as CR plus absence of phenotypically aberrant PCs (clonal) in bone marrow with a minimum of 1 million total bone marrow cells analyzed by multiparametric flow cytometry (with 2 tubes of 8colors) PET/CT negativity is defined as the complete disappearance of any area of fluorodeoxyglucose (FDG) uptake, according to the International Myeloma Working Group (IMWG) criteria
Definition of prognostic factors, as assessed by Next Generation Sequencing (NGS) (MM-panel) | 5 years
  An NGS-based MM-panel will be employed to deeply characterize MM CD138+ clone(s) both at diagnosis and at time of first PD. MM-panel includes genes either most frequently involved in MM pathogenesis, or involved in drugs' mechanism of action. In addition, it includes Single nucleotide polymorphisms (SNPs) located in genomic regions frequently involved in Chromosomal numerical abnormality (CNAs) in MM, as well as immunoglobulin heavy chain gene (IgH). The MM-panel will allow the exploitation of either genes' variants, or CNAs or IgH translocations as prognostic factors correlated to progression. In addition, the eventual variation of Variants Allele Frequencies (VAFs), as described in the comparison between diagnostic and progression CD138+ samples, will allow the definition of different evolutionary trajectories. A stratification of patients will be performed according to the evolution patterns, and clinical correlations will be performed.

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospital Ostrava, Ostrava, Czechia
- General Hospital of Athens "Alexandra", Athens, Greece
- A.O.U. Maggiore della Carità di Novara, Novara, Italy

IPD SHARING:
Plan to Share IPD: No